CLINICAL TRIAL: NCT05143710
Title: The Features of Clinical Imaging, Disease Severity and Pregnancy Outcomes in Posterior Reversible Encephalopathy Syndrome With Preeclampsia or Eclampsia
Brief Title: The Clinical and Prognostic Features of PRES
Status: Completed | Type: Observational
Sponsor: Dunjin Chen (Other)
Responsible Party: Sponsor-Investigator, Dunjin Chen, Director of obstetrics, Guangzhou Medical University
Organization: Guangzhou Medical University (Other)
Other Study IDs: 2020M682675
Record Dates: First submitted 2021-11-10; First posted 2021-12-03 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Posterior Reversible Encephalopathy Syndrome; Pregnancy Outcomes; Preeclampsia; Eclampsia
MeSH Terms: conditions — Posterior Leukoencephalopathy Syndrome; Pre-Eclampsia; Eclampsia | interventions — Pressure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PRES in PE or E: patients diagnosed with PRES in PE or E
  Interventions: Diagnostic Test: PRES in PE or E

INTERVENTIONS:
Diagnostic Test: PRES in PE or E — patients diagnosed with posterior reversible encephalopathy syndrome with preeclampsia or eclampsia

SUMMARY:
The purpose of this study is to determine the features of clinical imaging, disease severity and pregnancy outcomes in posterior reversible encephalopathy syndrome with preeclampsia or eclampsia.

DETAILED DESCRIPTION:
The investigators retrospectively collected data (General information, clinical data, biochemical indicators, imaging features, and pregnancy outcome) from pregnant woman diagnosed with PRES with preeclampsia or eclampsia to analyze features of clinical imaging, disease severity and pregnancy outcomes during 2012 to 2021.Then, the investigators grouped all the patients into early onset group and late onset PE group according to gestational weeks to analyze differences of clinical imaging. Finally, the investigators grouped all the patients into good pregnancy outcomes group and poor pregnancy outcomes group according to diagnostic criteria, including the incidence of stillbirth and premature birth, to analyze differences of clinical imaging .

ELIGIBILITY:
Inclusion Criteria:

1. patients were diagnosed of PRES with PE or E
2. all patients provided written informed consent

Exclusion Criteria:

1. patients combined with other neurological disorders
2. patients combined with mental illness

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pregnant woman diagnosed with PRES with preeclampsia or eclampsia
Sampling Method: Non-Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
features of clinical imaging | Cranial Imaging was examined immediately at the onset of symptoms, such as s headaches, visual changes, seizures, consciousness impairment, mental disorders, and focal neurological deficits.
  The imaging features were described by their location including frontal, parietal, occipital, temporal, cerebellum, basal ganglia, brain stem, deep white matter and callosum, and 1 point was recorded for each location involved.
blood pressure(BP) | The BP of patients was obtained immediately at the onset of symptoms.
  hypertension：≥140/90mmHg
biochemical parameters | Biochemical indicators were collected within 1 week of the hospital stay.
  The PRES patients may have a lower level of serum albumin (﹤35g/L) ,and have a higher level of lactic dehydrogenase (﹥380U/L).
pregnancy outcomes | The pregnancy outcomes will record immediately when the patients deliver.
  The rates of stillbirth and premature birth (gestation less than 37 weeks) in PRES patients.
pregnancy outcomes | From day of admission until the day of discharge or date of death from any cause,whichever came first,assessed up to 1 year.
  The PRES patients may have longer time of hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Key Laboratory for Major Obstetric Diseases of Guangdong Province, The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, China